CLINICAL TRIAL: NCT00772512
Title: Subject- And Investigator-Blinded, Sponsor-Open, Randomized, Single-Dose, Placebo-Controlled, 3-Way Crossover Study To Study Effects Of PF-04802540 On Polysomnography Endpoints In Healthy Volunteers
Brief Title: A Study Of The Effect Of PF-04802540 On Sleep Measures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taisho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B0911003
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: PF-04802540, polysomnography, REM, cross over

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: PF-04802540
- B (Experimental)
  Interventions: Drug: PF-04802540
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04802540 — 5 mg capsule, single dose
  Arms: A
Drug: PF-04802540 — 15 mg capsule, single dose
  Arms: B
Drug: Placebo — Placebo capsule, single dose
  Arms: C

SUMMARY:
The purpose of this study is to determine if PF-04802540 decreases REM sleep.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (nonchildbearing potential) subjects between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) between 18 to 32 kg/m2, inclusive, and a total body weight >45 kg (99 lbs)
* Non-users of nicotine

Exclusion Criteria:

* Evidence or history of clinically significant medical illness
* A history of seizures, including childhood febrile seizures
* Any condition possibly affecting drug absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
REM sleep percentage | 1 day

SECONDARY OUTCOMES:
REM sleep latency | 1 day
Beta EEG power | 1 day
Plasma concentrations of PF-04802540 and its metabolite, PF-04831035 | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New York, New York, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0911003&StudyName=A%20Study%20Of%20The%20Effect%20Of%20PF-04802540%20On%20Sleep%20Measures